CLINICAL TRIAL: NCT04788758
Title: Feasibility of Implementation and Assessment of Geriatric Assessment Screening Tool in Outpatient Oncology Clinic
Brief Title: Geriatric Assessment Screening Tool for the Identification of At-Risk Older Adults Who Are Undergoing Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19E.925; JT 14176 (Other: JeffTrial Number)
Record Dates: First submitted 2021-02-10; First posted 2021-03-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (G8 screening tool, referral) (Experimental): PHASE I: Registered Nurses receive training on how to administer the G8 screening tool utilizing an Epic flowsheet to patients using a self-directed education module and by direct assessment by a geriatrician.
  PHASE II: Patients complete the G8 screening tool questionnaire over 10 minutes as part of their standard initial assessment, and their answers are entered into their EHR flowsheet. Patients who score =< 14 on the G8 are referred for a CGA at SAOC, and these patients and their medical oncologists are made aware. Within 2 weeks of the initial screening, the results are communicated with the patient and medical oncologist at a 2-hour SAOC visit. Patients with a score of > 15 on the G8 are made aware of their results without any referral generated.
  Interventions: Other: Educational Intervention; Other: Screening Questionnaire Administration; Other: Referral; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive G8 screening tool administration training
  Other Names: Education for Intervention, Intervention by Education, Intervention through Education, Intervention, Educational
Other: Screening Questionnaire Administration — Complete G8 screening tool
Other: Referral — Receive referral
  Other Names: Referral, referral, Referred
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial investigates how easy it is to incorporate a nursing led geriatric assessment screening tool into a busy oncology practice, in order to identify at-risk older adults being evaluated for cancer treatment. This screening tool may help identify at-risk patients who can be referred for more in depth assessment, allowing for the creation of an individualized treatment plan that puts the patient's safety and personal goals as a priority.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of training nurses to administer the Geriatric 8 (G8) screening tool in an oncology practice, to identify older patients (> 65 years old [y/o]) that would benefit from a more extensive Comprehensive Geriatric Assessment (CGA).

SECONDARY OBJECTIVE:

I. To report the positive predictive value of the G8 screening tool with the final frailty designation determined by the Comprehensive Geriatric Assessment completed in patients referred to the Senior Adult Oncology Center (SAOC).

OUTLINE:

PHASE I:

Registered Nurses receive training on how to administer the G8 screening tool utilizing an Epic flowsheet to patients using a self-directed education module and by direct assessment by a geriatrician.

PHASE II:

Patients complete the G8 screening tool questionnaire over 10 minutes as part of their standard initial assessment, and their answers are entered into their electronic health record (EHR) flowsheet. Patients who score =< 14 on the G8 are referred for a CGA at SAOC, and these patients and their medical oncologists are made aware. Within 2 weeks of the initial screening, the results are communicated with the patient and medical oncologist at a 2-hour SAOC visit. Patients with a score of > 15 on the G8 are made aware of their results without any referral generated.

ELIGIBILITY:
Inclusion Criteria:

* NURSES: Assigned to two designated cancer clinics at Sidney Kimmel Cancer Center (SKCC) Center City, the Renal Cell Carcinoma (RCC) and Lymphoma/myeloma clinics
* PATIENTS: 65 years and older
* PATIENTS: Diagnosis of cancer

Exclusion Criteria:

• PATIENTS: Inability to answer or have caregiver answer questions on screening tool

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Overall assessment score: Pre | Before self-administered learning module
  The score will be a number between 1-20. The responses to two questions of primary interest, assessing their comfort caring for older adults and their comfort in administering the G8 tool, will be binary measurements. The overall assessment scores from pre- and post- self-administered learning module will be compared using paired Wilcoxon test.
Overall assessment score: Post | After self-administered learning module
  The score will be a number between 1-20. The responses to two questions of primary interest, assessing their comfort caring for older adults and their comfort in administering the G8 tool, will be binary measurements. The overall assessment scores from pre- and post- self-administered learning module will be compared using paired Wilcoxon test.
Number of patients screened | Up to 30 months
  Will be summarized by sample means, standard deviations and/or percentages.
Number of patients who refused | Up to 30 months
  Will be summarized by sample means, standard deviations and/or percentages.
Time it took to screen | Up to 30 months
  Will be summarized by sample means, standard deviations and/or percentages.
Number of referrals to Senior Adult Oncology Center (SAOC) | Up to 30 months
  Will be summarized by sample means, standard deviations and/or percentages.
Number of completed SAOC visits | Up to 30 months
  Will be summarized by sample means, standard deviations and/or percentages.

SECONDARY OUTCOMES:
Positive predictive value of the G8 | Up to 30 months
  The percentage of patients being determined as vulnerable/frail by Comprehensive Geriatric Assessment (CGA) at SAOC, i.e. the predictive positive value of G8, will be reported with its 95% confidence interval. The summary statistics of additional collected SAOC metrics including the Timed Up and Go test, prior history of falls, cognitive screen, depression screen, mortality prognostication, expected life expectancy, social distress thermometer, Mini Nutritional Assessment (MNA), presence of polypharmacy and inappropriate medications, and Eastern Cooperative Oncology Group (ECOG) score will be reported by means, standard deviations and percentages.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefefrson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No